CLINICAL TRIAL: NCT04312750
Title: An Open Label, Single-treatment, Single-period, Single-application, Adhesion Performance Study of Lidocaine Patch 36 mg/Patch (1.8%) in Healthy, Adult, Human Subjects.
Brief Title: Adhesion of Lidocaine Topical System 1.8%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCI-LIDO-ADH-001
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lidocaine Patch (Experimental): All subjects received one lidocaine topical system, which was applied to a predetermined fixed area on subject's left side of the back or right side of the back (lower/mid back) according to randomization schedule and worn for 12 hours.
  Interventions: Drug: Lidocaine topical system 1.8%

INTERVENTIONS:
Drug: Lidocaine topical system 1.8%
  Other Names: Lidocaine patch 1.8%; ZTlido

SUMMARY:
The objective of this study is to evaluate the adhesion performance of ZTlido (lidocaine topical system) 1.8% in normal, healthy volunteers.

DETAILED DESCRIPTION:
In this open-label, single-treatment, single-period, single-application adhesion performance study, 54 healthy, adult male and female subjects are treated with one lidocaine topical system to their back for 12 hours. Adhesion will be monitored throughout the wear time and skin irritation will be assessed after the topical system is removed.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on by medical history, laboratory work, and physical exam
* Be at least 18 years of age
* If childbearing potential, use of acceptable form of birth control
* In the case of females of childbearing potential, have a negative serum pregnancy test

Key Exclusion Criteria:

* Allergy or known hypersensitivity to lidocaine, amide-type local anesthetics, or any component of the product formulation
* Any major medical illness 3 months prior or any significant history or ongoing chronic medical illness
* Subjects with conditions that might affect application of the product or its adhesive properties (including psoriasis, eczema, atopic dermatitis, damaged or irritated epidermal layer, and excessive hair or oil on the skin)
* History of addiction, abuse, and misuse of any drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean Cumulative Adhesion Score | 0, 3, 6, 9, 12 hours post-dose
  Adhesion of the topical system to the skin is assessed by FDA 0-4 scoring system. The scoring for adhesion of topical systems is indicated as follows: 0 = ≥ 90% Adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% Adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% Adhered (less than half of the patch lifting off the skin), > 0% to < 50% Adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely detached). The mean cumulative adhesion score is calculated as the sum of scores at each assessment time point divided by the total number of observations.

SECONDARY OUTCOMES:
Dermal Response Score | 12.5 and 14 hours post-dose
  Product tolerability is assessed by Dermal Response Score. The application site is evaluated 30 minutes and 2 hours after product removal (12.5 and 14 hours post-dose, respectively). Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test (i.e., application) site.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Godfrey, PharmD, Principal Investigator — AXIS Clinicals

REFERENCES:
- [Derived] Gudin J, Webster LR, Greuber E, Vought K, Patel K, Kuritzky L. Open-Label Adhesion Performance Studies of a New Lidocaine Topical System 1.8% versus Lidocaine Patches 5% and Lidocaine Medicated Plaster 5% in Healthy Subjects. J Pain Res. 2021 Feb 23;14:513-526. doi: 10.2147/JPR.S287153. eCollection 2021. PMID 33654425